CLINICAL TRIAL: NCT05988853
Title: Efficacy of a Disinfection Protocol for Musical Instruments of a Music Therapy Service in Intensive Care Units
Brief Title: Biosafety of Musical Instruments in the ICU
Status: Completed | Type: Observational
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Mark Ettenberger, Coordinator Music Therapy Service, Fundación Santa Fe de Bogota
Other Study IDs: MTBIOSAFETY01
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Nosocomial Infection
Keywords: music therapy; biosafety; musical instruments; intensive care units
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: follow-up of patients — Follow-up of evidence of nosocomial infections of patients in music therapy

SUMMARY:
This study investigates the efficacy of the institutional disinfection protocol for musical instruments in the ICU of the music therapy service of the University Hospital Fundación Santa Fe de Bogotá (FSFB), Colombia.

DETAILED DESCRIPTION:
Introduction: Nosocomial infections can negatively affect the recovery and well-being of patients. Music therapy is a profession that uses music and sounds to improve the health, well-being and quality of life of patients. Musical instruments are regularly used in music therapy sessions, such as the string or percussion instruments, among others. Since the musical instruments are also played and handled by the patients, the question arises if the disinfection and cleaning protocol for musical instruments of the music therapy service at the University Hospital Fundación Santa Fe de Bogotá (FSFB) is effective and safe.

Objectives: To establish the effectiveness and impact of the disinfection protocol of musical instruments used by the music therapy service in the ICUs of the FSFB.

Methodology: This is a study carried out in 2 phases. The first phase corresponds to an experimental design in which the presence of microbiological viability will be evaluated through ATP bioluminescence tests and cultures before and after the application of the disinfection and cleaning protocol in a controlled environment. The second phase corresponds to a prospective cohort study in which music therapy patients will be followed up ver a period of two months, determining the impact of the disinfection and cleaning protocol.

Analysis: A descriptive analysis will be applied where the qualitative variables will be presented in their absolute and relative frequencies. For the quantitative variables, the Kolgomorov-Smirnov test will be applied to define the distribution of the data and, according to these, corresponding descriptive statistics will be carried out. In addition, a bivariate analysis will be performed between the outcome variable (infection or not) versus the exposure variables with a regression-type confounding analysis (logistic - binary as applicable) to identify co-variability phenomena.

Expected results: This study seeks to improve patient safety, raise awareness in the music therapy community about the importance of proper cleaning of their work tools, and promote inter- and transdisciplinary knowledge between the fields of music therapy, critical medicine and epidemiology.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized in the and having participated in a music therapy service from July 1st to August 31st 2023.

Exclusion Criteria:

* Not having participated in a music therapy service during the same time frame.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients hospitalized that have been part of the music therapy service from July 1st to August 31st 2023.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
ATP bioluminescence tests | 2 months
  ATP bioluminescence detects the amount of ATP, which is an indirect measurement of the amount of organic residue on a surface that has the potential to support microbial growth and also microbial biomass.
Microbial cultures | 2 months
  Will be taken if the ATP is positive (USP 42 <61>) or at least 10 microbial cultures will be taken randomly from the musical instruments used in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request.

REFERENCES:
- [Derived] Ettenberger M, Salgado A, Maya R, Merchan-Restrepo A, Barrera-Lopez P. Efficacy and Impact of a Cleaning and Disinfection Protocol for Musical Instruments Used in Music Therapy Services in ICUs: A Prospective Cohort Study. Jt Comm J Qual Patient Saf. 2024 Nov;50(11):755-763. doi: 10.1016/j.jcjq.2024.07.007. Epub 2024 Jul 26. PMID 39277481